CLINICAL TRIAL: NCT03275363
Title: The University of Hong Kong Neurocognitive Disorder Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Dementias Platform UK (Unknown)
Responsible Party: Principal Investigator, Dr Joseph SK Kwan, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: HKUNCDC
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Neurocognitive Disorder; Mild Cognitive Impairment; Alzheimer Dementia; Vascular Dementia; Age-related Cognitive Decline
Keywords: Subjective cognitive decline; Mild Cognitive Impairment; Dementia; Cerebral aging
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular; Dementia | interventions — Hematologic Tests; Electroencephalography; Evoked Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Venous blood at baseline and at yearly follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cognitively normal controls (CNC): No subjective memory complaints Normal HK-MoCA Normal instrumental ADL All interventions as described
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: MRI; Biological: Blood tests; Diagnostic Test: EEG with event-related potential (ERP)
- Subjective cognitive decline (SCD): Subjective memory complaints Normal HK-MoCA Normal instrumental ADL All interventions as described
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: MRI; Biological: Blood tests; Diagnostic Test: EEG with event-related potential (ERP); Diagnostic Test: Amyloid PET CT
- Mild cognitive impairment (MCI): Subjective memory complaints Low HK-MoCA Normal instrumental ADL All interventions as described
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: MRI; Biological: Blood tests; Diagnostic Test: EEG with event-related potential (ERP); Diagnostic Test: Amyloid PET CT
- Alzheimer's dementia: Subjective memory complaints Low HK-MoCA Poor instrumental ADL Probable Alzheimer's disease All interventions as described except EEG with ERP
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: MRI; Biological: Blood tests; Diagnostic Test: Amyloid PET CT
- Vascular dementia: Subjective memory complaints Low HK-MoCA Poor instrumental ADL Related to stroke / cerebrovascular disease All interventions as described except EEG with ERP
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: MRI; Biological: Blood tests; Diagnostic Test: Amyloid PET CT

INTERVENTIONS:
Diagnostic Test: Neurocognitive battery — Cognitive impairment status (SCD, MCI, dementia), HK-MoCA, Clinical Dementia Rating (CDR sum of squares), Geriatric Depression Scale (GDS-15), Neuropsychiatric Index (NPI), Barthel Index, Lawton's IADL, Life-Space Assessment, Mini-Nutrition Assessment (MNA), Quality of Life for Alzheimer's Disease (QoL-AD, patient and carer parts), frailty status (FRAIL scale), handgrip strength, walking speed, exercise status, sleep quality, Charlson comorbidity index (CCI, age-adjusted).
  NACC: Story recall, Benson's complex figure copy, colour trail test (black & white), verbal fluency, digit forward and backward span.
Diagnostic Test: MRI — MRI: T1, T2, FLAIR, SWI, DTI, fMRI, ASL, MRS, for selected patients
Biological: Blood tests — Stored samples (unanalysed): serum, plasma, buffy coat (PBMC); also processed for microvesicles and exosome analysis
Diagnostic Test: EEG with event-related potential (ERP) — 128-channel EEG with ERP for Go/NoGo and Prospective Memory (PM) tasks for selected patients
  Groups: Cognitively normal controls (CNC); Mild cognitive impairment (MCI); Subjective cognitive decline (SCD)
Diagnostic Test: Amyloid PET CT — F18 Flutametamol PET CT for selected patients
  Groups: Alzheimer's dementia; Mild cognitive impairment (MCI); Subjective cognitive decline (SCD); Vascular dementia

SUMMARY:
The HKU Neurocognitive Disorder (NCD) Cohort is a hospital-based, prospective, observational study of older HK Chinese adults with cognitive impairment, with a special focus on studying patients with subjective cognitive decline and mild cognitive impairment.

DETAILED DESCRIPTION:
The HKU Neurocognitive Disorder (NCD) Cohort is a hospital-based, prospective, observational study of older HK Chinese adults with cognitive impairment, with a special focus on studying patients with subjective cognitive decline and mild cognitive impairment, and in particular the biomarkers that predict cognitive and functional decline.

Comprehensive profiling of each subject is performed through a multi-domain assessment protocol including detailed demographics, lifestyle factors, neuropsychological battery, mood, MRI, genetics, blood biomarkers, and other patient-centred parameters including level of disability, quality of life and societal engagement. Ongoing annual follow up captures the essential clinical events and changes in neurocognitive function (conversion to MCI or dementia), mood, level of disability and quality of life; as well as repeat blood tests.

The HKU NCD Cohort is the first-ever Asian dementia cohort to be formally included into the Dementia Platforms UK, achieving an international collaborative status with other UK-based cohorts. The study neuropsychological battery is aligned with the NACC UDS3 battery.

ELIGIBILITY:
Inclusion Criteria:

* Older adults with or without neurocognitive disoder. HKU NCD Cohort focuses primarily on people with Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI).

Exclusion Criteria:

* Severe Parkinson's disease, major depressive disorder or severe psychiatric conditions, significant communication difficulties (e.g. aphasia, deafness), terminal cancer or likely end-of-life in the next 12 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults with or without neurocognitive disoder. HKU NCD Cohort focuses primarily on people with Subjective Cognitive Decline (SCD) and Mild Cognitive Impairment (MCI).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline | 1 year
  Change in total HK-MoCA score between baseline and follow-up

SECONDARY OUTCOMES:
Functional decline | 1 year
  Change in Lawton's IADL score between baseline and follow-up
Neuropsychiatric decline | 1 year
  Change in Neuropsychiatric Index (NPI) between baseline and follow-up
Quality of life decline | 1 year
  Change in QoL-AD score between baseline and follow-up
Change in cognitive impairment status | 1 year
  Progression to mild cognitive impairment (MCI) or dementia status

CONTACTS AND LOCATIONS:
Overall Officials: Joseph SK Kwan, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Share with Dementias Platform UK (www.dementiasplatform.uk)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Due to be shared from 2017, indefinitely.
Access Criteria: Via Dementias Platform UK (www.dementiasplatform.uk)
URL: http://www.dementiasplatform.uk